CLINICAL TRIAL: NCT00101491
Title: Partnership Programs to Reduce Cardiovascular Disparities - Deep South Partnerships for Prevention of CVD Disparities
Brief Title: STORIES-Stories to Communicate Risk About Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Catarina Kiefe, MD, PhD, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1282; U01HL079153 (NIH); U01HL079171 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Health Communication DVD video
- 2 (Other): Attention Control Comparator
  Interventions: Behavioral: Health Communication DVD video

INTERVENTIONS:
Behavioral: Health Communication DVD video — Interactive, testimonial-based, stage of change-matched Health Communication DVD video interventions

SUMMARY:
The purpose of this study is to develop and test an intervention based on literacy-appropriate electronic tools, tailored to the demographics and readiness for change of the user, to promote tobacco smoking cessation in a low-literacy population.

DETAILED DESCRIPTION:
PROJECT STORIES:

STORIES is one of two intervention trials conducted as part of the "Deep South Partnership for the Prevention of CVD Disparities" under the NHLBI Partnership Programs to Reduce Cardiovascular Disparities. STORIES is an innovative approach to smoking cessation programs provided in medical facilities for patients seeking assistance with quitting smoking. Our approach is to provide the patient with counseling prior to being discharged from the hospital in an effort to assist them with quitting smoking. The DVD will include current and previous smokers telling their stories regarding their tobacco use. We feel having the patient see other people similar to them express their views, struggles and successes with quitting smoking will motivate them to quit smoking. The patient will also receive 3 follow up telephone calls to check on their progress. Our hypothesis is that patients exposed to the interactive DVD will be more likely to quit, compared with those not exposed. The specific aims for this health communication project are: (1) to develop a series of interactive, testimonial-base stage of change-matched Health Communication DVD video interventions targeted at low-income, low-literacy African Americans in the Deep South and a health information interactive DVD for the patients selected in the randomized control group; (2) to train a peer health counselor/research assistant to counsel inpatient smokers to quit and assist the community members with learning to use the DVDs and then to follow-up by telephone at two weeks, three months and six months after discharge following enrollment in the project; and (3) to evaluate the impact of the intervention on processes of change and six month cessation rates among smokers using a group-randomized controlled trial.

The study completion date listed in this record was obtained from the "End Date" entered in the Query View Report (QVR) record.

ELIGIBILITY:
African American inpatients receiving treatment in the medicine unit who desire to quit smoking.

Inclusion Criteria:

* African Americans
* Patients not previously video/interviewed talking about smoking and health
* Patients willing to provide contact information for follow up
* Patients that are able to hear, view and communicate their input on material

Exclusion Criteria:

* Patients other than African American
* Admitted with issues of alcohol, drugs, and mentally unstable
* Patients leaving the state after hospitalization
* Patients without contact information for follow up
* Patients below age 19
* Non smokers
* Patients that use chewing tobacco
* Patients that are incarcerated

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | Measured at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Hullett, MD, MPH, Principal Investigator — Cooper Green Hospital; Catarina Kiefe, MD, PhD, Principal Investigator — University of Alabama at Birmingham; Thomas K Houston, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Cooper Green Hospital, Birmingham, Alabama
  - University of Alabama, Birmingham, Alabama

REFERENCES:
- [Derived] Cherrington A, Williams JH, Foster PP, Coley HL, Kohler C, Allison JJ, Kiefe CI, Volkman JE, Houston TK. Narratives to enhance smoking cessation interventions among African-American smokers, the ACCE project. BMC Res Notes. 2015 Oct 14;8:567. doi: 10.1186/s13104-015-1513-1. PMID 26467316
- See also: Alabama Collaboration for Cardiovascular Equality (ACCE) is an initiative under the leadership of Drs. Catarina Kiefe and Sandral Hullett and is comprised of STORIES (NCT00101491), led by Dr. Thomas Houston, and ADAPT (NCT00621569), led by Dr. Jamy Ard. — http://clinicaltrials.gov/show/NCT00621569